CLINICAL TRIAL: NCT02706756
Title: Conservative Intervention of Femoroacetabular Impingement Syndrome: A Randomized Controlled Trial
Brief Title: Conservative Intervention of Femoroacetabular Impingement Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar studies already published by other researchers
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00069234
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-02

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Musculoskeletal Manipulations; Exercise; Educational Status; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Education, exercise and manual therapy (Experimental): One group will receive education and advice, manual therapy that is applied toward the impairments of the subject, a prescription of progressive rehabilitation exercises designed to strengthen weakened muscle groups and stretch joint movements that demonstrate range of motion limitations. Treatment is based on clinical presentation and identification of impairments by the treating clinician. Subjects will be seen twice weekly for 4 to 6 weeks, depending on the progression.
  All three groups will receive standardized education on the current state of FAI interventions (with both conservative and surgical care). All interventions will be provided by licensed physical therapists that are named as investigators in this study.
  Interventions: Other: Manual therapy; Other: Education and advice
- Education and exercise (Active Comparator): Group will receive a prescriptive intervention designed to strengthen the hip and surrounding regions as well as improve flexibility of the lower extremity. This group will not receive additional physiotherapy management but will be schedule bi-weekly to review the home exercises and to receive appropriate educational support.
  All three groups will receive standardized education on the current state of FAI interventions (with both conservative and surgical care). All interventions will be provided by licensed physical therapists that are named as investigators in this study.
  Interventions: Other: Exercise; Other: Education and advice
- Supervised neglect (Placebo Comparator): Group will receive supervised neglect. We will monitor this group for changes or emergent situations but no formal care will be provided.
  All three groups will receive standardized education on the current state of FAI interventions (with both conservative and surgical care). All interventions will be provided by licensed physical therapists that are named as investigators in this study.
  Interventions: Other: Education and advice; Other: Supervised neglect

INTERVENTIONS:
Other: Manual therapy — Hip joint and spine manual therapy techniques applied toward the impairments of the subject.
  Arms: Education, exercise and manual therapy
Other: Exercise — Prescriptive exercise program of self-mobilization and/or strengthening program to address impairments of the subject.
  Arms: Education and exercise
Other: Education and advice — All three groups will receive standardized education on the current state of FAI interventions (with both conservative and surgical care).
Other: Supervised neglect — Monitoring of group without formal intervention.
  Arms: Supervised neglect

SUMMARY:
1. Purpose: 1) compare three conservative treatment approaches for subjects with femoroacetabular impingement syndrome (FAI), and 2) analyze functional outcome comparatively across groups.
2. Interventions will be provided based on randomized assignment. Group 1 will receive treatment based on identified impairments and treated twice weekly to address said impairments with hip manual therapy and exercise, as well as a prescriptive exercise for strengthening and mobility of the hip. Group 2 will receive only the prescriptive exercise program. Group 3 will be a control group (supervised neglect)
3. Primary outcomes data analysis will involve a mixed design (repeated measures) ANOVA for assessment of the primary outcome measure of the HAGOS. Secondary analyses will include chi square analyses (PASS, surgery at 6 months, adverse events), ANCOVA (PPMs, and expectations measures), or other appropriate comparative measures. None of the proposed treatment is considered outside of 'standard of practice'.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 18 to 60 years,
* diagnosed with FAI by an orthopedic surgeon and exhibiting
* hip/groin symptoms for at least 3 months (symptomatic); and
* signs, symptoms and imaging findings conducive to FAI will be recruited from a surgical practice of an orthopedic surgeon in Durham, North Carolina.

Exclusion Criteria:

* subjects that have radiographic evidence of hip osteoarthritis that is more than mild in severity defined as Tonnis >grade 1 or Kellgren-Lawrence >2;
* have other concurrent injury/conditions that will affect their ability to participate in the rehabilitation program and/or assessment procedures;
* exhibit hip dysplasia (center edge angle <20 degrees on AP radiograph
* are unable to attend a study physiotherapist or participate in the rehabilitation program if randomized to the PT group;
* are unable to understand English.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Did subject elect to undergo surgery? | up to 6 months after intervention
  Determination of whether the subject had surgery for femoroacetabular impingement or not

SECONDARY OUTCOMES:
Change in Stanford Expectations of Treatment Scale (SETS) | initial visit, 4 to 6 weeks after initial visit, and 6 months after initial visit
  subject expectation of treatment
Change in Patient Acceptable Symptom State (PASS) | initial visit, 4 to 6 weeks after initial visit, and 6 months after initial visit
  subject acceptance of what their current symptom state is
Change in numeric pain rating scale | initial visit, 4 to 6 weeks after initial visit, and 6 months after initial visit
Change in Hip and Groin Outcome Score | initial visit, 4 to 6 weeks after initial visit, and 6 months after initial visit
Change in Single leg stance (SLS) | initial visit, 4 to 6 weeks after initial visit, and 6 months after initial visit
  measure of single leg balance and stability
Change in Lower Quarter Y Balance Test (YBT-LQ) | initial visit, 4 to 6 weeks after initial visit, and 6 months after initial visit
  measure of single leg balance, strength and coordination
Change in Single Leg Anteroposterior Hop | initial visit, 4 to 6 weeks after initial visit, and 6 months after initial visit
  Measure of single leg balance, strength, power and coordination
Change in Standing Hip Internal Rotation Range-of-Motion | initial visit, 4 to 6 weeks after initial visit, and 6 months after initial visit
  Measure of single leg weight-bearing range of motion
Change in Complications/Adverse Events of assigned treatment | initial visit, 4 to 6 weeks after initial visit, and 6 months after initial visit

IPD SHARING:
Plan to Share IPD: No